CLINICAL TRIAL: NCT06628284
Title: Dexcom CGM as Preventative Diagnostic Tool in Steroid-Induced Hyperglycemia During Interventional Pain Management Procedure
Brief Title: CGM as Diagnostic Tool in Observing Steroid-Induced Hyperglycemia
Acronym: TRC-DX-1
Status: Completed | Type: Observational
Sponsor: Mahesh Pattabiraman (Industry)
Responsible Party: Sponsor-Investigator, Mahesh Pattabiraman, Chief Executive, TriCity Research Center
Organization: TriCity Research Center (Industry)
Other Study IDs: IIS-23-DEX-001
Record Dates: First submitted 2024-09-29; First posted 2024-10-04 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Diabetes; Pain Management
MeSH Terms: conditions — Diabetes Mellitus; Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Test Group: The study will be conducted as a single-arm trial consisting of participants enrolled in the test group. Each participant will receive a G7 CGM and their blood glucose levels will be continuously transmitted to the Dexcom Clarity cloud system for monitoring and data collection.
  Interventions: Device: Dexcom G7

INTERVENTIONS:
Device: Dexcom G7 — The study will be conducted as a single-arm trial consisting of participants enrolled in the test group. Each participant will receive a G7 CGM and their blood glucose levels will be continuously transmitted to the Dexcom Clarity system for monitoring and data collection. As a observational study, the test group glucose levels will be monitored after receiving a steroid for pain management. The CGM profile of steroid-induced hyperglycemia in patients will be studied for the following corticosteroids: dexamethasone (10 mg), methylprednisolone (40 mg or 80 mg), triamcinolone (40 mg or 80 mg).

SUMMARY:
This study is designed to help understand how certain steroid medications affect blood sugar levels in patients undergoing pain management treatments. Patients who receive steroid injections for conditions like back pain or arthritis experience temporary high blood sugar (called steroid-induced hyperglycemia, SIH), which can sometimes lead to complications, especially in patients with diabetes. This study aims to understand this by monitoring blood glucose levels using continuous glucose monitors (Dexcom G7). The main goal of this study is to track how steroid injections impact blood sugar levels in patients.

DETAILED DESCRIPTION:
Steroid injections are frequently used in pain management for conditions such as arthritis, back pain, and joint inflammation. While effective at reducing pain and inflammation, these steroids can cause temporary spikes in blood sugar, known as steroid-induced hyperglycemia. This can be a concern, especially for patients with diabetes, as poorly managed high blood sugar can lead to serious complications. This study aims to explore the effects of three commonly used steroids: dexamethasone, methylprednisolone, and triamcinolone, each administered at different doses. Participants will be fitted with a Dexcom G7 continuous glucose monitor (CGM) on their arm, which will track their blood sugar levels every 5 minutes for up to 10 days.

The study's primary objective is to determine how often steroid-induced hyperglycemia occurs, how severe it is, and how long it lasts. Study will also investigate whether certain factors-such as the type of steroid, dosage, or the patient's underlying conditions-affect blood sugar responses. Additionally, the study will assess how the use of the CGM device may improve overall patient care, reduce the need for emergency interventions, and potentially lower healthcare costs by preventing complications.

By gathering high-resolution glucose data, this research will provide valuable insights into the best practices for managing blood sugar in patients receiving steroid injections. Our goal is to improve treatment strategies, particularly for diabetic patients, ensuring safer and more effective pain management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19-75 years
* Patients meeting the medical criteria for need of interventional pain management procedure requiring corticosteroid administration.
* Willing and able to use Dexcom's CGM device.
* Willing to install Dexcom G7 app in their phone and register it for cloud data sharing
* Able to understand and sign informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Medically unmanaged diabetes
* History of diabetic ketoacidosis (DKA) or hyperosmolar hyperglycemic state (HHS)
* History of severe hypoglycemia
* Active infection
* History of a liver disorder (ALT > threefold of the ULN)
* History of any renal disease
* Immune compromised patient
* Active illegal drug user (self-reported)
* Under any other steroid treatment
* Any other medical condition or treatment that would make participation in the study unsafe or infeasible.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult participants aged 19-75 years who are undergoing interventional pain management procedures requiring corticosteroid administration. Participants must be willing and able to use the Dexcom G7 Continuous Glucose Monitoring system and install the corresponding app on their smartphones. Eligible participants must meet the medical criteria for corticosteroid use in pain management, as determined by the principal investigator, and must provide informed consent prior to participation. Exclusion criteria include pregnancy, medically unmanaged diabetes, history of severe hypoglycemia or diabetic ketoacidosis, active infections, or any conditions that would make the study unsafe or infeasible as determined by the investigator
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Spike in blood glucose level (hyperglycemic phase) | From baseline (day 0) to end of monitoring (day 10)
  Hyperglycemic phase is determined based on clinically significant increase in percentage points above baseline
Duration of hypo- or hyperglycemia | From baseline (day 0) to end of monitoring (day 10)
  minutes of blood glucose level in hypo-/hyperglycemic phase
Drop in blood glucose levels (hypoglycemic phase) | From baseline (day 0) to end of monitoring (day 10)
  Hypoglycemic phase is determined based on clinically significant decrease in percentage points below baseline

SECONDARY OUTCOMES:
Hospitalization rates | From baseline (day 0) to end of monitoring (day 10)
  Electronic health record analysis
Number of phone calls to study team | From baseline (day 0) to end of monitoring (day 10)
  Analysis of electronic health records

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Grand Island Pain Relief Center, Grand Island, Nebraska
  - Hastings Pain Relief Center, Hastings, Nebraska

IPD SHARING:
Plan to Share IPD: Undecided
The research team is open to sharing individual participant data with qualified researchers who meet the appropriate criteria for data access. However, the team may decide against sharing due to concerns about the sensitive nature of the glucose monitoring data, the potential risks of re-identification even with anonymized datasets, and the need to protect patient confidentiality. Additionally, data governance and patient consent considerations may also influence the decision to withhold IPD sharing.